CLINICAL TRIAL: NCT01014364
Title: Phase III Study of Hydrocortisone in Patients With Severe H1N1 Related Pneumonia
Brief Title: Low Doses Corticosteroids as Adjuvant Therapy for the Treatment of Severe H1N1 Flu
Acronym: CORTIFLU
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: the H1N1 pandemic is now over, and fewer cases than expected were observed
Sponsor: University of Versailles (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Djillali Annane, Dean of the health Science Centre, University of Versailles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCR09006
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Pneumonia, Viral; Influenza in Humans
Keywords: Acute lung injury; Acute respiratory distress syndrome; corticosteroids; inflammation
MeSH Terms: conditions — Pneumonia, Viral; Influenza, Human; Acute Lung Injury; Respiratory Distress Syndrome; Inflammation | interventions — Hydrocortisone; hydrocortisone acetate; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Corticosteroids (Experimental): Hydrocortisone
  Interventions: Drug: hydrocortisone
- Control (Placebo Comparator): isotonic saline
  Interventions: Drug: isotonic saline

INTERVENTIONS:
Drug: hydrocortisone — 50mg intravenous bolus every 6 hours for one week, then every 12 hours for one week and then every 24 hours for one week
  Other Names: hydrocortisone acetate
  Arms: Corticosteroids
Drug: isotonic saline — intravenous bolus every 6 hours for one week, then every 12 hours for one week and then every 24 hours for one week
  Other Names: normal saline
  Arms: Control

SUMMARY:
The H1N1 flu pandemic is one of the major infectious threat of the past half century. it is rapidly progressing worldwide and a substantial number of patients get severe H1N1 related pneumonia that requires mechanical ventilation and admission to the intensive care unit. The acute respiratory distress syndrome is associated with a substantial mortality and morbidity partly as a consequence of uncontrolled lung and systemic inflammation. many physicians are trying to counteract this pro-inflammatory storm by the use of corticosteroids albeit these drugs may cause super infection or metabolic disorders. Thus, there is a need for a randomized double blind, placebo controlled trial to define the benefit to risk ratio of corticosteroids in this patient.

ELIGIBILITY:
Inclusion Criteria:

* age above 15 years old
* admitted to intensive care unit
* proven or strong suspicion of H1N1 Influenza infection
* diffuse pneumonia (for less than 96 hours)
* need for non invasive or invasive mechanical ventilation

Exclusion Criteria:

* pregnancy
* an age of 15 or less
* rapidly fatal underlying disease with a life expectancy of one month or less
* more than 3 organ dysfunction upon admission
* previous treatment with corticosteroids (ie prednisone 30 mg per day or more, or equivalent, for at least one month)
* formal indication for corticosteroids (eg Addison disease, status asthmaticus)
* already on corticosteroids for 2 days or more in the management of the current episode
* acute lung injury not related to viral pneumonia
* presence of H1N1 related acute myocarditis or encephalitis
* receiving antiviral treatment for more than 5 days

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
in hospital all cause morality | hospital discharge up to 90 days

SECONDARY OUTCOMES:
28 day mortality | 28 day
90 day all cause mortality | 90 day
6 month all cause mortality | 180 days
mechanical ventilation free days | hospital discharge up to 90 days
intensive care unit free days | hospital discharge up to 90 days
proportion of patients with secondary infections | hospital discharge up to 90 days
proportion of patients who require ECMO | hospital discharge up to 90 days
respiratory function and health status | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Djillali Annane, MD,PhD, Study Chair — AP--HP and University of Versailles SQY; Christian Brun Buisson, MD, Principal Investigator — AP-HP and Paris XII University; Charles Mayaud, Principal Investigator — AP-HP and University of Paris VII; Bernard Régnier, Principal Investigator — AP-HP and Paris VII University; Christian Perronne, Principal Investigator — AP-HP and University of Versailles SQY
Locations (1):
- Raymond Poincaré hospital, Garches, France

REFERENCES:
- [Result] Annane D, Antona M, Lehmann B, Kedzia C, Chevret S; CORTIFLU Investigators; CRICs; AZUREA; REVA/SRLF networks. Designing and conducting a randomized trial for pandemic critical illness: the 2009 H1N1 influenza pandemic. Intensive Care Med. 2012 Jan;38(1):29-39. doi: 10.1007/s00134-011-2409-8. Epub 2011 Nov 26. PMID 22120766